CLINICAL TRIAL: NCT07075809
Title: The Effectiveness of Laserpuncture on Chemotherapy-induced Leucopenia and Quality of Life in Head and Neck Cancer Patients
Brief Title: The Effectiveness of Laserpuncture on Chemotherapy-induced Leucopenia in Head and Neck Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Resti Victoria Fanggidae, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 25-06-0942
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Leucopenia Induced Chemoteraphy Adult

STUDY DESIGN:
Intervention Model Description: the laser acupuncture will be designated as the investigation group while the sham laser acupuncture will be designated as the control group
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participants and the outcome assessors will be blinded to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigation Group (Experimental): The laser acupuncture
  Interventions: Device: The laser acupuncture
- Control Group (Sham Comparator): The sham laser acupuncture
  Interventions: Device: Sham Laser acupuncture

INTERVENTIONS:
Device: The laser acupuncture — The intervention group in this study receives laser acupuncture therapy using a laser Micropad GL2+ device with an infrared wavelength of 880 nm. The laser acupuncture is applied to specific acupuncture points, namely GV14, LI4, ST36, and SP6 on the body, as well as ear points including MA-TF1 Shenmen, MA-SC5 Liver, MA-IC3 Endocrine, MA-IC8 Spleen, and MA-SC6 Kidney. Treatment is administered once daily for a total of six sessions during the chemotherapy treatment period.
  Arms: Investigation Group
Device: Sham Laser acupuncture — The Control group in this study receives sham laser acupuncture therapy using a laser Micropad GL2+ device with deactivation mode. The sham laser acupuncture is applied to specific acupuncture points, namely GV14, LI4, ST36, and SP6 on the body, as well as ear points including MA-TF1 Shenmen, MA-SC5 Liver, MA-IC3 Endocrine, MA-IC8 Spleen, and MA-SC6 Kidney. Treatment is administered once daily for a total of six sessions during the chemotherapy treatment period.
  Arms: Control Group

SUMMARY:
The goal of this clinical trial is to evaluate if laserpuncture (laser acupuncture) can reduce leucopenia caused by chemotherapy and improve the quality of life in patients with head and neck cancer. The main questions it aims to answer are:

* Does laserpuncture reduce the incidence of chemotherapy-induced Leucopenia ?
* Does laserpuncture improve quality of life in these patients?

Researchers will compare patients receiving laserpuncture therapy to a control group receiving sham laserpuncture to see if the intervention has a beneficial effect.

Participants will:

* Undergo six sessions of laserpunktur or sham laserpuncture during chemotherapy
* Have leukocyte counts and absolute neutrophil counts measured before and 7-14 days after chemotherapy
* Complete quality of life assessments using EORTC QLQ-C30 and EORTC QLQ-H&N35 questionnaires

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with head and neck cancer, aged 18-60 years.
* Head and neck cancer patients diagnosed through histopathological examination, with cancer stages II to IV.
* Head and neck cancer patients undergoing chemotherapy with platinum-based chemotherapy drugs combined with 5-Fluorouracil, in the first treatment cycle.
* Leukocyte count greater than 5000/mm³.
* Patients who have signed informed consent and are willing to participate in the study until completion.
* Normal Mini-Mental State Examination (MMSE) score (27-31).

Exclusion Criteria:

* Patients with cancer lesions, ulcers, acute dermatitis, or exacerbation of chronic skin diseases at the selected acupuncture points.
* Patients with deformities or anatomical abnormalities of the ear.
* Patients with fever (body temperature >38ºC).
* Patients with hemodynamic instability (patient vital signs outside the normal limits. Normal vital signs include axillary temperature of 36.5 - 37.5ºC, systolic blood pressure 102 - 131 mmHg, diastolic blood pressure 61 - 83 mmHg, pulse rate 60 - 100 beats/minute. Unstable if respiratory rate is above 25 breaths/minute or SpO2 < 90%).

Patients with a history of allergy to laser irradiation (skin hypersensitivity due to exposure to specific light).

- Patients with a history of uncontrolled seizures or epilepsy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2025-10-01 (Actual); Primary Completion 2025-12-12 (Actual); Study Completion 2025-12-12 (Actual)

PRIMARY OUTCOMES:
Leukocyte Count | Before therapy, between 7-14 day after chemoterapy
  Leukocyte count is the measure of the number of white blood cells (leukocytes) present in the blood
Absolute Neutrophil Count | Before therapy, between 7-14 day after chemoterapy
  The Absolute Neutrophil Count (ANC) is a laboratory measure of the number of neutrophils, a type of white blood cell that plays a critical role in fighting infection, present in the blood.
European Organization of Research and Treatment of Cancer Quality of Life Questionnaire- Core 30 questionnaire | Before therapy, between 7-14 day after chemoterapy
  Self-reported questionnaire to assess the quality of life of cancer patients.
European Organization of Research and Treatment of Cancer Quality of Life Questionnaire Heand &Neck 35 questionnaire | Before therapy, between 7-14 day after chemoterapy
  Self-reported questionnaire to assess quality of life specific to patients with head and neck cancer.

CONTACTS AND LOCATIONS:
Overall Officials: KPEK FKUI-RSCM, Principal Investigator — The Health Research Ethics Commitee of Faculty of Medicine
Locations (1):
- Universitas Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided